CLINICAL TRIAL: NCT03458871
Title: Home Neuromodulation of the Neurogenic Bladder in Chronic Spinal Cord Injury With Transcutaneous Tibial Nerve Stimulation
Acronym: HomeTTNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Argyrios Stampas, MD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0423
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Results first posted 2020-03-04 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Spinal Cord Injury; Neurogenic Bowel
Keywords: electric stimulation
MeSH Terms: conditions — Neurogenic Bowel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 4-week TTNS home based protocol (Experimental): Transcutaneous Tibial Nerve Stimulation (TTNS) applied to subjects for 4-week protocol.
  Interventions: Device: 4-week TTNS home-based protocol

INTERVENTIONS:
Device: 4-week TTNS home-based protocol — 4-week TTNS home-based protocol. Electrodes 2 inch by 2 inch will be placed according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is not contraction seen, maximal tolerable intensity will be used.
  In addition, if the patient perceives pain, the intensity will be lowered until comfortable.
  Stimulation frequency of 10 Hz and pulse width of 200ms in continuous mode will be used.

SUMMARY:
Determine the safety, feasibility, compliance, and efficacy of a daily home TTNS protocol in chronic SCI provided by self or caregiver for 4 weeks.

DETAILED DESCRIPTION:
In Specific Aim 1, we will monitor for safety, feasibility, and compliance of a home TTNS program for bladder management. In Specific Aim 2, the efficacy of home TTNS will be compared to baseline Incontinence- Quality of Life questionnaire. A bladder diary will also capture important information such as frequency and volume of catheterization, incontinence episodes, and other related observations.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Neurologically stable SCI for ≥ 6 months
* Intermittent catheterization to empty bladder
* Stable bladder medications for ≥ 3 months

Exclusion Criteria:

* Multiple medications for the bladder
* Other diagnoses to explain incontinence (ex: UTI, bladder stones, multiple sclerosis, etc.)
* 2+ pitting edema that does not resolve
* Known peripheral neuropathy or injury to the path of the tibial nerve
* Demand-type cardiac pacemaker or implanted defibrillator
* Cancer in the tibial nerve path and/or bladder
* Inability to elicit toe/plantar flexion with electric stimulation during the clinic visit.
* Inability to understand directions
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Argyrios Stampas, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Stampas A, Korupolu R, Lee KH, Salazar B, Khavari R. Reduction of Overactive Bladder Medications in Spinal Cord Injury With Self-Administered Neuromodulation: A Randomized Trial. J Urol. 2024 Dec;212(6):800-810. doi: 10.1097/JU.0000000000004189. Epub 2024 Aug 2. PMID 39093916

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-week TTNS Home Based Protocol: Transcutaneous Tibial Nerve Stimulation (TTNS) applied to subjects for 4-week protocol.
  4-week TTNS home-based protocol: 4-week TTNS home-based protocol. Electrodes 2 inch by 2 inch will be placed according to anatomic landmarks, with the negative electrode behind the internal malleolus and the positive electrode 10cm superior to the negative electrode, verified with rhythmic flexion of the toes secondary to stimulation of the flexor digitorum and hallicus brevis. The intensity level will be set to the amperage immediately under the threshold for motor contraction. If there is not contraction seen, maximal tolerable intensity will be used.
  In addition, if the patient perceives pain, the intensity will be lowered until comfortable.
  Stimulation frequency of 10 Hz and pulse width of 200ms in continuous mode will be used.
Period: Overall Study
Arm/Group | 4-week TTNS Home Based Protocol
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 2
  Hispanic | 6
  White | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Years of injury [Median (Inter-Quartile Range); unit: years] | 8.75 [3.1 to 19.4]
Number of participants on bladder medication [Count of Participants; unit: Participants] | 14
American Spinal Injury Association Impairment Scale Level [Count of Participants; unit: Participants] — The ASIA Scale has four levels of impairment, as follows: AIS A= complete injury; AIS B= motor complete injury; AIS C= motor incomplete injury with less than half of muscles below the motor level with antigravity strength; and AIS D= motor incomplete injury with at least half of the muscles below the motor level with antigravity strength.
  Participants
    A | 11
    B | 2
    C | 2
    D | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Using TTNS at Home Daily as Indicated by Number of Adverse Events Recorded in Bladder Diary
Description: Noted on bladder diary will be description of observed changes including but not limited to pain, fatigue, vision changes, mental status, bowel program changes, and sexual function changes. The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 1
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Number; unit: adverse events
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
adverse events | 0

2. Primary Outcome: Safety of Using TTNS at Home Daily as Indicated by Number of Adverse Events Recorded in Bladder Diary
Description: Noted on bladder diary will be description of observed changes, including but not limited to pain, fatigue, vision changes, mental status, bowel program changes, and sexual function changes. The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 2
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Number; unit: adverse events
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
adverse events | 0

3. Primary Outcome: Safety of Using TTNS at Home Daily as Indicated by Number of Adverse Events Recorded in Bladder Diary
Description: as for outcome 2
Time Frame: week 3
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Number; unit: adverse events
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
adverse events | 1

4. Primary Outcome: Safety of Using TTNS at Home Daily as Indicated by Number of Adverse Events Recorded in Bladder Diary
Description: as for outcome 2
Time Frame: week 4
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Number; unit: adverse events
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
adverse events | 1

5. Primary Outcome: Compliance as Assessed by Number of Days Per Week TTNS Was Used, as Recorded at Home Daily in Bladder Diary
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 1
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
days | 6.9 (0.5)

6. Primary Outcome: Compliance as Assessed by Number of Days Per Week TTNS Was Used, as Recorded at Home Daily in Bladder Diary
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 2
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
days | 7 (0)

7. Primary Outcome: Compliance as Assessed by Number of Days Per Week TTNS Was Used, as Recorded at Home Daily in Bladder Diary
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 3
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
days | 7 (0)

8. Primary Outcome: Compliance as Assessed by Number of Days Per Week TTNS Was Used, as Recorded at Home Daily in Bladder Diary
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 4
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
days | 6.6 (1.3)

9. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 1
Population: This data was not collected.
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 0

10. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 2
Population: This data was not collected.
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 0

11. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 3
Population: This data was not collected.
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 0

12. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "TTNS Was Easy to Use"
Description: The TTNS satisfaction survey ranges from 0 (strongly disagree) to 10 (strongly agree), with higher scores indicating greater satisfaction.
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 9.4 (1.7)

13. Secondary Outcome: Quality of Life as Assessed by Score on Incontinence of Quality of Life (I-QOL) Survey
Description: Total score on the I-QOL survey is reported. The total score ranges from 0 (poor quality of life) to 100 (maximum quality of life), with a higher score indicating a better quality of life.
Time Frame: week 0
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 55.6 (4.67)

14. Secondary Outcome: Quality of Life as Assessed by Score on Incontinence of Quality of Life (I-QOL) Survey
Description: as for outcome 13
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 70.2 (17.0)

15. Secondary Outcome: Quality of Life as Assessed by Score on Incontinence of Quality of Life (I-QOL) Survey
Description: as for outcome 13
Time Frame: week 4
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 59.1 (3.51)

16. Secondary Outcome: Number of Catheterizations Per Day
Description: Frequency of catheterization after TTNS. The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 1, week 2, week 3, week 4
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: catherizations per day
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
catherizations per day
  week 1 | 5.2 (1.7)
  week 2 | 5.1 (1.8)
  week 3 | 5.4 (1.8)
  week 4 | 5.4 (2)

17. Secondary Outcome: Volume of Catheterization
Description: The research assistant will call weekly to capture the written data and monitor progress with the protocol.
Time Frame: week 1, week 2, week 3, week 4
Population: Only 14 of the 16 participants used the bladder diary, which was used to collect this data.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 14
milliliters
  week 1 | 366 (131.4)
  week 2 | 332 (129.6)
  week 3 | 340.1 (140.2)
  week 4 | 342.6 (138.9)

18. Secondary Outcome: Anticholinergic Side Effect Severity as Assessed by an Anticholinergic Side Effect Severity of Symptom Questionnaire
Description: Items on the anticholinergic side effect severity of symptom questionnaire is scored as 0 (None), 1 (Mild), 2 (Moderate), or 3 (Severe), with a higher score indicating a worse outcome.
Time Frame: week 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale
  Dry Mouth | 1.00 (1.15)
  Constipation | 0.50 (0.97)
  Hard Stool | 0.75 (0.77)
  Sleepy | 1.06 (0.93)
  Decreased Cognition | 0.25 (0.58)

19. Secondary Outcome: Anticholinergic Side Effect Severity as Assessed by an Anticholinergic Side Effect Severity of Symptom Questionnaire
Description: as for outcome 18
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale
  Dry Mouth | 0.38 (0.62)
  Constipation | 0.44 (0.81)
  Hard Stool | 0.38 (0.72)
  Sleepy | 0.56 (0.81)
  Decreased Cognition | 0.19 (0.54)

20. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "It Was Not Embarrassing to Use TTNS"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 9.375 (2.420)

21. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "It Was Easy to Remember to Use TTNS"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 9.875 (0.484)

22. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "TTNS Did Not Irritate my Skin"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 9.375 (2.420)

23. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "TTNS Was Not Painful"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 10 (0)

24. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "TTNS Improved my Quality of Life"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 5.6 (3.9)

25. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "I Enjoyed Using TTNS"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 8.3 (3.5)

26. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "If TTNS Works as Well as Medications, I Would Switch to TTNS"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 8.4 (3.5)

27. Primary Outcome: Overall Satisfaction of Daily Use of TTNS at Home as Assessed by a TTNS Satisfaction Survey - Item "Overall, I Would Recommend TTNS for Those With Neurogenic Bladder"
Description: as for outcome 12
Time Frame: week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week TTNS Home Based Protocol
Number analyzed (Participants) | 16
score on a scale | 9.7 (1.3)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | 4-week TTNS Home Based Protocol
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4-week TTNS Home Based Protocol (N=16)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT03458871/Prot_SAP_000.pdf